CLINICAL TRIAL: NCT01688804
Title: A Mobile Health Approach to Reducing Sedentary Time in Bariatric Surgery Patients
Brief Title: Reducing Sedentary Time in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R03DK095740-01 (NIH)
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2012-09

CONDITIONS: Sedentary Behavior
Keywords: Sedentary behavior; Physical activity; Obesity; Mobile health; Smartphone
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral intervention (Experimental): Behavioral intervention to reduce sedentary time delivered via mobile smartphone
  Interventions: Behavioral: Behavioral intervention to reduce sedentary time delivered via mobile smartphone

INTERVENTIONS:
Behavioral: Behavioral intervention to reduce sedentary time delivered via mobile smartphone — The overall goals of the intervention are to decrease overall sedentary time and to increase the number of breaks in sedentary time. The intervention approach combines an advanced smartphone device with an on-board accelerometer and a sophisticated smartphone application to: 1) monitor participants sedentary behavior in real time in their natural environment; and 2) use monitored data to deliver immediate, individually-tailored, goal-driven prompts and feedback to encourage substitute of sedentary behaviors with physical activity.

SUMMARY:
Greater time spent in sedentary behaviors, independent of physical activity level, can increase risk of morbidity and mortality. Objective assessments indicate that bariatric surgery patients spend large amounts of time in sedentary behaviors. The present study is the first to test whether a mobile health (mHealth) approach that employs widely adopted smartphone technology to monitor and modify sedentary behaviors as they occur is a feasible and acceptable method of reducing sedentary time in these patients and other obese populations.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery patients and other obese individuals will be considered
* Body mass index >= 30 kg/m2

Exclusion Criteria:

* Report being unable to engage in daily activities and walk continuously for >= 10 minutes without assistance
* Are currently involved in a physical activity intervention.
* Are unable to read or understand the study materials
* Are currently taking medications that cause dizziness and/or feeling faint when sitting or standing.
* Report any condition that in the opinion of investigators would preclude adherence to the intervention protocol including plans to relocate, history of substance abuse or other significant psychiatric problems, or terminal illness.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Average daily sedentary minutes | 4 weeks

SECONDARY OUTCOMES:
Average daily adherence to prompts to reduce sedentary time delivered via mobile smartphone | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dale S Bond, Ph.D., Principal Investigator — The Miriam Hospital/Brown Alpert Medical School
Locations (1):
- The Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Bond DS, Thomas JG, Raynor HA, Moon J, Sieling J, Trautvetter J, Leblond T, Wing RR. B-MOBILE--a smartphone-based intervention to reduce sedentary time in overweight/obese individuals: a within-subjects experimental trial. PLoS One. 2014 Jun 25;9(6):e100821. doi: 10.1371/journal.pone.0100821. eCollection 2014. PMID 24964010
- See also: Related Info — http://www.weightresearch.org/fundedgrants.html